CLINICAL TRIAL: NCT03362203
Title: The Hypersensitivity and Changes of Conditioned Pain Modulation in Chronic Neck Pain Patients
Brief Title: Conditioned Pain Modulation in Chronic Neck Pain Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, guochen, Department of Spine Surgery, Peking University People's Hospital
Other Study IDs: Neckpainspine001
Record Dates: First submitted 2017-11-26; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Neck Pain
Keywords: Conditioned pain modulation, neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with chronic neck pain: Patients,aged 21-80 years, must have experienced neck pain for at least 3 months and have reported a minimal pain level of 30 (pain threshold) on the 0-100 pain numerical rating scale (NRS) in the last 7 days.
  Interventions: Other: Patients with chronic neck pain
- Subjects without chronic neck pain: Subjects,aged 21-80 years, must not have presented episodes of chronic neck pain for more than 7 days in the last 12 months.
  Interventions: Other: Subjects without chronic neck pain

INTERVENTIONS:
Other: Patients with chronic neck pain — Patients,aged 21-80 years, must have experienced neck pain for at least 3 months and have reported a minimal pain level of 30 (pain threshold) on the 0-100 pain numerical rating scale (NRS) in the last 7 days.
  Groups: Patients with chronic neck pain
Other: Subjects without chronic neck pain — Subjects,aged 21-80 years, must not have presented episodes of chronic neck pain for more than 7 days in the last 12 months.
  Groups: Subjects without chronic neck pain

SUMMARY:
The aim of this study was to evaluate changes in local and segmental hypersensitivity and endogenous pain inhibition in people with chronic nonspecific neck pain.

DETAILED DESCRIPTION:
Quantitative sensory testing is widely used in human research to investigate the state of the peripheral and central nervous system contributions in pain processing. It is a valuable tool to help identify central sensitization and may be important in the treatment of chronic neck pain. This study is a cross-sectional study. Two groups including chronic neck pain group and healthy volunteers group will be arranged in this study. The healthy subjects will be matched for sex and age in relation to the neck pain group. The pressure pain threshold (PPT) will be measured at the neck muscle in both groups. The cold pressor test will be used in both groups to activate conditioned pain modulation.

ELIGIBILITY:
1. Chronic neck pain subjects

   Inclusion criteria:
   * Age 21-80 years old.
   * People must have experienced neck pain for at least 3 months and have reported a minimal pain level of 30 (pain threshold) on the 0-100 pain numerical rating scale (NRS) in the last 7 days.

   Exclusion Criteria:
   * Age under 21 or over 80.
   * Patients were excluded if they had taken pain medications on the day of the assessment or if they had serious spinal pathologies, such as fractures, tumors or inflammatory diseases, such as ankylosing spondylitis, nerve root compromise confirmed by clinical neurological tests or severe cardiorespiratory diseases.
   * Those who were pregnant, patients with cancer and those with a cardiac pacemaker were also excluded.
2. Healthy volunteers

Inclusion criteria:

* Age 21-80 years old.
* These participants must not have presented episodes of low back pain for more than 7 days in the last 12 months.

Exclusion Criteria:

* Age below 21 or over 80 years old.
* These participants have presented episodes of low back pain for more than 7 days in the last 12 months.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Chronic neck pain subjects People must have experienced neck pain for at least 3 months and have reported a minimal pain level of 30 (pain threshold) on the 0-100 pain numerical rating scale (NRS) in the last 7 days.Patients were excluded if they had taken pain medications on the day of the assessment or if they had serious spinal pathologies. Those who were pregnant, patients with cancer and those with a cardiac pacemaker were also excluded.
  2. Healthy volunteers These participants must not have presented episodes of low back pain for more than 7 days in the last 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
Change of pressure pain threshold (PPT) | The PPT will be measured before CPT, 30 seconds after the CPT begin, and immediately after CPT.
  A cold pressor test (CPT) was used to induce pain and trigger the conditioned pain modulation (CPM) response. The conditioned stimulus was immersion of the leg in a bucket of ice water on the side ipsilateral to the most painful neck region. The neck PPT was recorded beginning 30 s after immersion of the leg with two PPT measures for each point. The PPT will be also measured again immediately after CPT.

SECONDARY OUTCOMES:
Numerical rating scale for pain (NRS) | The patients used this scale to rate the pain intensity of the neck pain before the experiment.
  The NRS evaluates levels of pain intensity using an 100-point scale (range 0-100), with 0 being classified as "no sensation", 30 "pain threshold", 100 "pain as bad as could be".

CONTACTS AND LOCATIONS:
Overall Officials: Chen Guo, Master, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dailey DL, Rakel BA, Vance CGT, Liebano RE, Amrit AS, Bush HM, Lee KS, Lee JE, Sluka KA. Transcutaneous electrical nerve stimulation reduces pain, fatigue and hyperalgesia while restoring central inhibition in primary fibromyalgia. Pain. 2013 Nov;154(11):2554-2562. doi: 10.1016/j.pain.2013.07.043. Epub 2013 Jul 27. PMID 23900134
- [Background] Xia W, Morch CD, Matre D, Andersen OK. Exploration of conditioned pain modulation effect on long-term potentiation-like pain amplification in humans. Eur J Pain. 2017 Apr;21(4):645-657. doi: 10.1002/ejp.968. Epub 2016 Oct 20. PMID 27766711
- [Background] Neziri AY, Dickenmann M, Scaramozzino P, Andersen OK, Arendt-Nielsen L, Dickenson AH, Curatolo M. Effect of intravenous tropisetron on modulation of pain and central hypersensitivity in chronic low back pain patients. Pain. 2012 Feb;153(2):311-318. doi: 10.1016/j.pain.2011.10.008. Epub 2011 Nov 17. PMID 22100357